CLINICAL TRIAL: NCT02136199
Title: Patient-centered Dissemination of Evidence-based Medicine: Share EBM
Brief Title: Use of Decision Aids in Clinical Encounters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Victor Montori, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 14-002055
Record Dates: First submitted 2014-03-24; First posted 2014-05-12 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Diabetes, Depression, Cardiovascular Disease,Hypercholesterolemia, Osteoporosis
MeSH Terms: conditions — Diabetes Mellitus; Depression; Cardiovascular Diseases; Hypercholesterolemia; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Implementation of Share EBM Toolkit (Other): Investigators led implementation of tailored activities and tactics (Shared EBM Toolkit) designed to promote the use of the decision aids in clinical encounters (i.e. journal clubs, value map streaming).
  Interventions: Other: Active Implementation of ShareEBM Toolkit
- Passive Implementation of Share EBM Toolkit (Other): Locally supported dissemination of Shared EBM Toolkit designed to promote the use of the decision aids in clinical encounters.
  Interventions: Other: Passive Dissemination of Share EBM

INTERVENTIONS:
Other: Active Implementation of ShareEBM Toolkit
  Arms: Active Implementation of Share EBM Toolkit
Other: Passive Dissemination of Share EBM
  Arms: Passive Implementation of Share EBM Toolkit

SUMMARY:
The active strategy for dissemination and implementation of Share Evidence Based Medicine (EBM) will yield greater reach of clinicians, be adopted by the practices more readily, and a greater uptake of use amongst encounters will be seen.

The Institute for Clinical Systems Improvement (ICSI) is a nonprofit organization with expertise in large-scale practice improvement at the state and national level. Largely funded by health organizations in Minnesota, ICSI has a sustainable model to translate evidence into practice, through clinical practice guidelines, shared decision making, and practice redesign. A partnership between these two organizations (ICSI and Mayo Clinic) may lead to a sustainable and innovative approach to the dissemination of evidence-based health information at the point of care.

The objective of the current study is therefore to leverage the expertise of these two organizations to compare the impact of an active to a passive dissemination and implementation strategy of the ShareEBM toolkit. The aim of the study is to disseminate evidence-based information through the use of decision aids during encounters. The overall purpose of the qualitative evaluation is to understand why decision aids were used more or less in certain practices and what factors contributed to or hindered this uptake.

ELIGIBILITY:
Inclusion Criteria:

* Practices meeting the following criteria will be deemed eligible for the study if they have:

  1. At least 2 primary care clinicians committed to participate in the study. Clinicians are defined as any healthcare professional providing patient care (i.e., physicians, nurse practitioners, physician assistants, diabetes educators)
  2. A designated site champion and support staff that can provide the support needed to conduct the study
  3. An IRB approval from their institution or are covered under Mayo Clinic IRB
  4. Leadership is committed to this research and has endorsed the study
* Any clinician caring for patients with a chronic condition and who has opportunities to discuss medication management with their patients will be deemed eligible

Exclusion Criteria:

* Major barriers to participating or to providing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of use of decision aids in clinical encounters by weekly reports | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Victor Montori, MD, Principal Investigator — Mayo Clinic
Locations (12):
- United States (12):
  - Park Nicollet- Brookdale, Brooklyn Center, Minnesota
  - Ridgeview Medical Center, Delano, Minnesota
  - Essentia Health-Lakeside Clinic, Duluth, Minnesota
  - Fairview Clinic-Eagan, Eagan, Minnesota
  - Park Nicollet-Golden Valley, Golden Valley, Minnesota
  - Essentia Hermantown Clinic, Hermantown, Minnesota
  - Native American Community Clinic, Minneapolis, Minnesota
  - Community Health Service, Inc., Rochester, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Fairview Medical-Rosemount, Rosemount, Minnesota
  - Baldwin Area Medical Center, Inc., Baldwin, Wisconsin
  - Hudson Physicians S.C., Hudson, Wisconsin